CLINICAL TRIAL: NCT06031584
Title: A Phase Ib/II Clinical Study to Evaluate the Safety and Efficacy of BL-M07D1 for Injection in Patients With Locally Advanced or Metastatic HER2-positive/Low-expressing Urinary and Gastrointestinal Solid Tumors
Brief Title: A Study of BL-M07D1 in Patients With a Variety of Solid Tumors Including Locally Advanced or Metastatic HER2-positive/Low-expressing Urinary and Gastrointestinal Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-202
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Her2-positive/Low-expression Urinary and Digestive Tract Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants received BL-M07D1 therapy in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-M07D1

INTERVENTIONS:
Drug: BL-M07D1 — BL-M07D1 was administered by intravenous infusion every 3 weeks in 3-week cycles.

SUMMARY:
Phase Ib: Explore the safety and tolerability of BL-M07D1 to further define RP2D in a variety of solid tumors, including locally advanced or metastatic urinary and gastrointestinal tumors. Phase II: To explore the efficacy of BL-M07D1 in patients with a variety of solid tumors including locally advanced or metastatic HER2-positive/low-expressing urinary and gastrointestinal tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Patients with unresectable locally advanced or metastatic HER2-positive/low-expressing urological and digestive system tumors, as well as other solid tumors;
6. Agree to provide archived tumor tissue specimens or fresh tissue samples from primary or metastatic lesions within the past 2 years;
7. Must have at least one measurable lesion as defined by RECIST v1.1;
8. ECOG performance status score of 0 or 1;
9. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50%;
11. Organ function levels must meet the requirements;
12. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
13. Urine protein ≤2+ or ≤1000 mg/24h;
14. Albumin ≥30 g/L;
15. For premenopausal women with childbearing potential, a pregnancy test (serum/urine) must be performed within 7 days before starting treatment, and the result must be negative; they must not be breastfeeding. All enrolled patients (regardless of gender) must use adequate barrier contraception throughout the treatment period and for 7 months after treatment ends.

Exclusion Criteria:

1. Received chemotherapy, biological therapy, immunotherapy, or other antitumor treatments within 4 weeks or 5 half-lives prior to the first dose;
2. Previously treated with ADC drugs containing camptothecin derivatives as payloads;
3. History of severe cardiovascular or cerebrovascular diseases;
4. Active autoimmune or inflammatory diseases;
5. History of other malignancies within 5 years prior to the first dose;
6. Thrombotic events requiring therapeutic intervention within 6 months before screening;
7. Patients with significant pleural/peritoneal/pelvic effusion or pericardial effusion, or those with symptomatic effusion, or poorly controlled effusion;
8. Poorly controlled hypertension despite antihypertensive medication;
9. Current interstitial lung disease, drug-induced interstitial pneumonitis, radiation pneumonitis requiring steroid treatment, or history of these conditions;
10. Patients with primary central nervous system (CNS) tumors or CNS metastases that failed local treatment;
11. History of hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies, or any excipients of BL-M07D1;
12. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation;
13. Positive for human immunodeficiency virus (HIV) antibodies, active tuberculosis, or active hepatitis C virus (HCV) infection;
14. Active hepatitis B virus (HBV) infection (exclusion criterion);
15. Severe infection requiring systemic treatment within 4 weeks before the first dose of the study drug;
16. Participation in another clinical trial within 4 weeks before the first dose;
17. Pregnant or lactating women;
18. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study.
Phase II: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase Ib/II: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.
Phase Ib: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib/II: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib/II: Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase II: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Phase Ib/II: Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M07D1 will be investigated.
Phase Ib/II: Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M07D1 will be investigated.
Phase Ib: T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-M07D1 will be investigated.
Phase Ib: AUC0-t | Up to approximately 24 months
  Blood concentration - Area under time line.
Phase Ib: CL | Up to approximately 24 months
  The serum clearance rate of BL-M07D1 per unit time will be investigated.
Phase Ib/II: Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M07D1 prior to the next dose will be administered.
Phase Ib/II: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-BL-M07D1 antibody (ADA) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, PHD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China